CLINICAL TRIAL: NCT03895398
Title: Effectiveness of Post Disaster Nutrition Intervention to Optimize Growth and Development of Under-two-year-old Children in Lombok, Indonesia
Brief Title: Post Disaster Nutrition Intervention for Under-two-year-old Children in Lombok Indonesia
Acronym: NIELombok
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Collaborators: Indonesia-MoH (Other Government); Indonesia University (Other)
Responsible Party: Principal Investigator, Dr.Umi Fahmida, Principal Investigator, SEAMEO Regional Centre for Food and Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIELombok
Record Dates: First submitted 2019-02-23; First posted 2019-03-29 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Weight Gain
Keywords: underfive children; post-disaster recovery; optimized food based recommendation; growth; development; psycho-social stimulation
MeSH Terms: conditions — Weight Gain | interventions — Nutritional Status; Psychosocial Intervention

STUDY DESIGN:
Intervention Model Description: in the intervention arm: ECE teachesr, community health officers, mother, and children will received treatment in the form of trainings (for ECE teachers and community health officers), parenting class (for mother), and nutrient dense food supplementation (for children) whilst in the control arm will received nothing as comparison to the intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nutrition and psychosocial intervention arm (Experimental): 12 selected ECE centers will be selected to be the intervention group. ECE teachers will be trained on psychosocial and nutrition care for children and expected to deliver the information and parenting class to mother.
  Community health officers will be trained on how to monitored the activities regularly and providing technical assistance to ECE teachers if needed.
  mothers will received weekly parenting class. in the parenting class mothers will be informed on how to provide appropriate feeding and psychosocial stimulus to their children. nutrient dense food supplementation in the form of liver and fish floss will be prepared together and distributed.
  underfive children will received nutrient dense food supplementation in the form of liver and fish floss and expected to be eaten everyday for 6 months
  Interventions: Other: nutrition and psychosocial intervention with community participatory
- control arm (No Intervention): no intervention is given to this arm

INTERVENTIONS:
Other: nutrition and psychosocial intervention with community participatory — community participation to ensure the intervention is given to the study subject (underfive children)
  Arms: nutrition and psychosocial intervention arm

SUMMARY:
In 2018, multiple earthquake with magnitude range from 6 to 7 hit Lombok Island, West Nusa Tenggara Province, Indonesia. Following the situational analysis and baseline study in December 2018 (4 months after the first earthquake), it was found that the prevalence of wasting and underweight of underfive children in the affected population is moderate (10.2% and 28.8%) but the prevalence of stunting and anemia is considered of highly significant public health problem (33.3% and 43.8%). Various organizations have provided support at the emergency phase but there is no specific program for nutrition support at the rehabilitation phase.

Draft of intervention model which utilize early child education (ECE) centers as center of nutrition recovery in the community has been discussed with the local education and health officers. Training will be delivered to ECE teachers and community health officers. ECE teachers are expected to have regular parenting class for nutrition education and activities, whilst the community health officers will monitor the activities and provide technical guidance as needed. Mothers of the underfive children will be invited to attend weekly parenting class at nearby ECE center in which they receive messages related to infant and young child feeding (IYCF), including distribution of liver and fish floss as nutrient dense food supplement to their children, and provision of appropriate psychosocial care.This parenting class will be held for 6 months with regular monitoring from the researchers and health personnel from public health center. Effectiveness of the intervention will be assessed in improving IYCF practices and psychosocial care of mothers and nutrient intakes, nutritional status and developmental outcomes of the underfives children.

DETAILED DESCRIPTION:
This study aims to strengthen management of nutrition program during post-disaster recovery for underfive children. In this study the following steps will be carried out.

Phase 1: Situation analysis is carried out with two approaches. The first approach is to analyze secondary data in the form of data related to nutrition, health and description of the affected population. The second approach is primary data collection by conducting a qualitative study in the form of in-depth interviews and focus group discussion (FGD) involving the local government and other parties related to the disaster management in East Lombok. Then, interviews and FGDs will be conducted to chief of villages and staff, community leaders and refugees, especially mothers with children under five children to complete data on the status and IYCF practices. The results of this situation analysis will be reported to the local government and also used as a basis for improving the implementation of the next stage.

Phase 2: Preparation of technical guidelines for the nutrition recovery program for underfive children by the research team based on situation analysis and literature review which has been carried out previously.

Stage 3: Representatives from ECE teachers and health workers from Public Health Centers will be trained on the implementation of parenting class and its monitoring. Then, together with the researchers, ECE teachers and community health workers will carry out the weekly parenting class, periodic monitoring and program evaluation.

Stage 4: At this stage there will be an intervention in the form of nutrient-dense food supplementation and psychosocial care for mothers with the concept of "Community Participation". Mothers and community members such as cadres will be involved in joint activities to provide nutrient-dense food for underfives children.

Stage 5: At the end of the activity an evaluation and monitoring program will be conducted by the research team in collaboration with the district health office.

ELIGIBILITY:
Inclusion Criteria:

* age ranged between 6-13 months and 24-49 months
* live with their mother / main caregiver
* parents consent to join the study
* live in affected areas

Exclusion Criteria:

* has chronic / congenital diseases
* have sibling that already join the study

Ages: 6 Months to 49 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
nutritional status | 6 months of intervention
  weight gain in g/kg.day

SECONDARY OUTCOMES:
protein intake | 6 months of intervention
  protein intake (gram/day)
development | 6 months of intervention
  Bayley Scales of Infant Development (BSID) as total score (range 0 - >115)
psycho-social care | 6 months of intervention
  HOME Inventory score as total score (range 0-45)
iron intake | 6 months of intervention
  iron intake (mg/day)
zinc intake | 6 months of intervention
  zinc intake (mg/day)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Wangge, Study Chair — SEAMEO RECFON
Locations (1):
- Seameo Regional Center for Food and Nutrition, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Sioen GB, Sekiyama M, Terada T, Yokohari M. Post-Disaster Food and Nutrition from Urban Agriculture: A Self-Sufficiency Analysis of Nerima Ward, Tokyo. Int J Environ Res Public Health. 2017 Jul 10;14(7):748. doi: 10.3390/ijerph14070748. PMID 28698515
- [Background] Fahmida U, Santika O, Kolopaking R, Ferguson E. Complementary feeding recommendations based on locally available foods in Indonesia. Food Nutr Bull. 2014 Dec;35(4 Suppl):S174-9. doi: 10.1177/15648265140354S302. PMID 25639135
- See also: UNHCR Emergency Handbook REPORTfrom UN High Commissioner for Refugees Published on 12 Jun 2015 — https://reliefweb.int/report/world/unhcr-emergency-handbook